CLINICAL TRIAL: NCT01998633
Title: Reduced-Intensity Conditioning for Children and Adults With Hemophagocytic Syndromes or Selected Primary Immune Deficiencies (RICHI) (BMT CTN #1204)
Brief Title: Reduced Intensity Conditioning for Hemophagocytic Syndromes or Selected Primary Immune Deficiencies (BMT CTN 1204)
Acronym: RICHI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN1204; 2U10HL069294-11 (NIH); 5U24CA076518 (NIH)
Record Dates: First submitted 2013-10-29; First posted 2013-12-02 (Estimated); Results first posted 2018-06-01 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Hemophagocytic Lymphohistiocytosis; Chronic Active Epstein-Barr Virus Infection; Chronic Granulomatous Disease; HIGM-1; Leukocyte Adhesion Deficiency; IPEX
Keywords: Hemophagocytic lymphohistiocytosis; Chronic Active EBV; Chronic Granulomatous Disease; Hyperimmunoglobulin M Syndrome (Hyper IGM); Leukocyte Adhesion Deficiency; IPEX; Hematopoietic Stem Cell Transplant (HSCT); Non-Myeloablative Transplant (NST); Reduced-Intensity Conditioning (RIC)
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic; Granulomatous Disease, Chronic; Hyper-IgM Immunodeficiency Syndrome; Leukocyte adhesion deficiency type 1 | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hematopoietic Stem Cell Transplant (Experimental): Participants will undergo a non-myeloablative allogeneic hematopoietic stem cell transplant.
  Interventions: Biological: Hematopoietic Stem Cell Transplant

INTERVENTIONS:
Biological: Hematopoietic Stem Cell Transplant — NOTE: The - sign is the number of days before the transplant and the + sign is the number of days after the transplant.
  * Alemtuzumab 0.2mg/kg Day-14,-13,-12,-11,-10
  * Fludarabine 30 mg/m2 on Day -8,-7,-6,-5,-4
  * Melphalan 140mg/m2 on Day -3
  The GVHD prophylaxis will consist of the following:
  * Cyclosporine on Day -3 to Day +100, maintaining a level of 250-500 ng/mL, then taper to Day +180.
  * Methylprednisolone 2 mg/kg/day on Day -2 and -1, 1 mg/kg/day on Day 0 to Day +28, then taper over 1 month. Oral prednisone may be substituted starting on Day 0 (1.2 mg/kg/day)

SUMMARY:
HLH, HLH-related disorders, Chronic Granulomatous (CGD), HIGM1, Immune dysregulation, polyendocrinopathy, enteropathy, and X-linked inheritance (IPEX) and severe LAD-I represent primary immune disorders that are typically fatal without Hematopoietic Cell Transplant (HCT). However, transplant is often complicated by inflammation, infection and other co-morbidities. In addition, these disorders have been shown to be cured with partial chimerism, making them an ideal target for the use of reduced intensity approaches, where a portion of patients may not achieve full donor chimerism, but instead achieve stable mixed chimerism. Reduced-intensity conditioning strategies have demonstrated improved survival with decreased Treatment Related Mortality (TRM) in institutional series for patients with HLH (Cooper et al., 2006; Marsh et al., 2010; Marsh et al., 2011). However, graft loss and unstable chimerism remain challenges. An institutional case series from Cincinnati Children's Hospital demonstrated full or high-level chimerism and improved durable engraftment using intermediate (Day -14) timing alemtuzumab (Marsh et al., 2013b). This study aims to test the efficacy of the Intermediate RIC strategy in a prospective multi-center study including HLH as well as other primary immunodeficiencies where allogeneic transplant with RIC has been shown to be feasible and stable chimerism is curative.

DETAILED DESCRIPTION:
The primary goal of this Phase II clinical trial is to determine the one-year overall survival of patients treated for immune deficiencies including HLH, HLH-like disorders, CGD, HIGM1, IPEX syndrome, and severe LAD-I with Matched Related Donor (MRD)/ Matched Unrelated Donor (MUD) bone marrow transplant using a reduced-intensity conditioning strategy including intermediate-timing of alemtuzumab. The donor choice is an unaffected related bone marrow donor who is a 6/6 match at HLA-A, -B (intermediate or higher resolution) and -DRB1 (at high resolution using DNA-based typing) OR a 7/8 or 8/8 match for human leukocyte antigen (HLA)-A, -B, -C and -DRB1 (at high resolution using DNA-based typing), OR an unrelated bone marrow donor who is a 7/8 or 8/8 match at HLA-A, -B, -C and -DRB1 (at high resolution using DNA-based typing). The transplant conditioning regimen will include fludarabine, melphalan, and alemtuzumab starting at Day -14 (Flu/Mel/Alem). Graft Versus Host Disease (GVHD) prophylaxis will consist of cyclosporine and corticosteroids through engraftment. Post-transplant supportive care will include infection surveillance and prophylaxis, and disease-specific supportive care.

ELIGIBILITY:
Inclusion Criteria

1. Patient is ≥ 3 months and ≤ 45 years of age at time of enrollment.
2. Meets criteria for one of the following immune disorders (2A-2F) requiring HCT:

2A. HLH or related disorder with indication for HCT [a. Inherited gene mutation associated with HLH: PRF1, UNC13D (MUNC13-2), STXBP2 (MUNC18-2), STX11, RAB27A (Griscelli syndrome, type 2), SH2D1A (XLP1), XIAP (XLP2), LYST (Chediak-Higashi syndrome) - OR - b. Meets clinical criteria for HLH, refractory to therapy according to HLH-94 or HLH-2004 (dexamethasone/etoposide), or recurrent episodes of hyper-inflammation - OR - c. Meets clinical criteria for HLH, without identified gene defects, with affected sibling - OR - decreased or absent NK cell function at the last evaluation, - OR - a history of CNS inflammation as evidenced by pleocytosis in CSF or MRI evidence of hyper-inflammation in the CNS]

2B. CAEBV: Patients with chronic EBV infection (CAEBV) with or without associated lymphoma (in complete remission) or active HLH. Note that this diagnosis is distinct from post-transplant lymphoproliferative disorder/ EBV-associated lymphoproliferative disease (PTLD/LPD). [Patients must meet all of the following: a. Severe progressive illness, usually with fever, lymphadenopathy and splenomegaly that either began as primary EBV infection or was associated with markedly elevated antibody titers to EBV viral capsid antibody (≥ 1:5120) or early antigen (≥ 1:640), or markedly elevated EBV DNA in the blood; - AND - b. Infiltration of tissues (e.g., lymph nodes, liver, lungs, CNS, bone marrow, eye, skin) with lymphocytes; - AND - c. Elevated EBV DNA, RNA or proteins in affected tissues; - AND - d. The absence of HIV or post-transplant lymphoproliferative disorder]

2C. Chronic granulomatous disease with indication for HCT [a. Oxidative burst < 10% normal with dihydrorhodamine (DHR) assay - AND - b. Documented CGD mutation(s) in gp91phox, p47phox, p67phox, p22phox or p40phox - AND - c. Severe disease as evidenced by one or more of the following: history of one or more potentially life-threatening infections; inflammatory bowel disease; failure to thrive with height <10% for age (unless parent(s) height <10%); or autoimmune complication felt to be linked to CGD]

2D. X-linked Hyper IgM Syndrome (HIGM1) [a. Decreased serum IgG (more than 2 standard deviations below normal for age) - AND - b. Mutation in CD40LG - OR - family history of maternally related males with HIGM1]

2E. IPEX Syndrome [a. Absent FOXP3+ CD4+ T cells - OR - abnormal function of FOXP3+CD4+ T cells - AND - b. Disease-associated mutation in FoxP3 (bi-allelic in females) - OR - family history of maternally related males with clinical diagnosis of IPEX]

2F. Severe Leukocyte Adhesion Deficiency, type I (LAD-I) [a. Decreased CD18 expression on neutrophils (<5% normal for age) - AND - b. Mutation of ITGB2 - OR - absence of ITGB2 mRNA in leukocytes]

3. Lansky or Karnofsky performance status ≥ 50%.

4. The patient's donor must be willing and able to give bone marrow stem cells and be:

a. An unaffected sibling donor who is a 6/6 match at HLA-A and -B (intermediate or higher resolution) and -DRB1 (at high resolution using DNA-based typing) OR b. An unaffected related donor (other than sibling) who is a 7/8 or 8/8 match for HLA-A, -B, -C (at intermediate or higher resolution) and -DRB1 (at high resolution using DNA-based typing) OR c. An unrelated donor who is a 7/8 or 8/8 match at HLA-A, -B, -C, and -DRB1 (at high resolution using DNA-based typing).

5. Patient must have adequate organ function as measured by:

1. Cardiac: Left ventricular ejection fraction (LVEF) > 40%; or LV shortening fraction (LVSF) > 26% by echocardiogram.
2. Renal: Calculated or radioisotope Glomerular Filtration Rate (GFR) > 50 mL/min/1.73m^2
3. Hepatic: Adequate liver function: serum conjugated (direct) bilirubin < 2x upper limit of normal for age as per local laboratory (with the exceptions of isolated hyperbilirubinemia due to Gilbert's syndrome, or hyperbilirubinemia as the result of liver inflammation in the setting of persistent, active HLH); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 10x upper limit of normal as per local laboratory (with the exception of elevated transaminase levels as the result of liver inflammation in the setting of persistent, active HLH).
4. Pulmonary: Patient may not be on mechanical ventilation support or have progressive pulmonary infection at the time of transplant; Pulmonary Function Testing (PFT) with forced expiratory volume in one second (FEV1) > 50% of normal and Diffusing capacity of the lung for carbon monoxide (DLCO) corrected for Hgb > 50% of normal. Patients unable to undergo PFTs should have stable respiratory status with SaO2 > 90% on a maximum of 2L/min supplemental oxygen.

   6. Signed informed consent.

   Exclusion Criteria:
   1. Hematopoietic stem cell transplant within 6 months of enrollment.
   2. Uncontrolled bacterial, viral or fungal infection (currently receiving appropriate antimicrobials and experiencing progression or no clinical improvement) at time of enrollment. We recognize that patients with CAEBV may have ongoing EBV viremia at the time of initiating transplant therapy, but other patients should have no uncontrolled bacterial, viral or fungal infections at the time of enrollment (or prior to initiating the preparative regimen).
   3. Pregnant or breastfeeding.
   4. Seropositive for human immunodeficiency virus (HIV).
   5. Alemtuzumab within 2 weeks of enrollment.
   6. History of prior or current malignancy, especially malignancies with a likelihood of relapse and progression, with the exception of (1) EBV-associated lymphomas related to immune deficiency or lymphomas associated with X-linked LPD in a good remission, as they are unlikely to relapse after treatment; (2) Resected basal cell carcinoma or treated cervical carcinoma in situ. Cancer treated with curative intent will not be allowed unless approved by the Protocol Officer or one of the Protocol Chairs.

Ages: 4 Months to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-09-23 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, MS, Study Director — Center for International Blood and Marrow Transplant Research (CIBMTR), Medical College of Wisconsin
Locations (22):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins, Baltimore, Maryland
  - Dana Farber Cancer Institute/Children's Hospital of Boston, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Washington University/St. Louis Children's Hospital, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Medical Center of Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Midwest Children's Cancer, Milwaukee, Wisconsin
- Canada (3):
  - British Columbia Children's Hosp-Vancouver, Vancouver, British Columbia
  - Hopital Sainte-Justine, Montreal, Quebec
  - McGill University - Montreal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Findings will be published in a manuscript.
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public.
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Background] Przepiorka D, Weisdorf D, Martin P, Klingemann HG, Beatty P, Hows J, Thomas ED. 1994 Consensus Conference on Acute GVHD Grading. Bone Marrow Transplant. 1995 Jun;15(6):825-8. PMID 7581076
- [Background] Filipovich AH, Weisdorf D, Pavletic S, Socie G, Wingard JR, Lee SJ, Martin P, Chien J, Przepiorka D, Couriel D, Cowen EW, Dinndorf P, Farrell A, Hartzman R, Henslee-Downey J, Jacobsohn D, McDonald G, Mittleman B, Rizzo JD, Robinson M, Schubert M, Schultz K, Shulman H, Turner M, Vogelsang G, Flowers ME. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. Biol Blood Marrow Transplant. 2005 Dec;11(12):945-56. doi: 10.1016/j.bbmt.2005.09.004. PMID 16338616
- [Derived] Geerlinks AV, Scull B, Krupski C, Fleischmann R, Pulsipher MA, Eapen M, Connelly JA, Bollard CM, Pai SY, Duncan CN, Kean LS, Baker KS, Burroughs LM, Andolina JR, Shenoy S, Roehrs P, Hanna R, Talano JA, Schultz KR, Stenger EO, Lin H, Zoref-Lorenz A, McClain KL, Jordan MB, Man TK, Allen CE, Marsh RA. Alemtuzumab and CXCL9 levels predict likelihood of sustained engraftment after reduced-intensity conditioning HCT. Blood Adv. 2023 Jul 25;7(14):3725-3734. doi: 10.1182/bloodadvances.2022009478. PMID 37042921

RESULTS

PARTICIPANT FLOW:
Groups:
- Hematopoietic Stem Cell Transplant: Participants will undergo a non-myeloablative allogeneic hematopoietic stem cell transplant.
  Hematopoietic Stem Cell Transplant: NOTE: The - sign is the number of days before the transplant and the + sign is the number of days after the transplant.
  * Alemtuzumab 0.2mg/kg Day-14,-13,-12,-11,-10
  * Fludarabine 30 mg/m2 on Day -8,-7,-6,-5,-4
  * Melphalan 140mg/m2 on Day -3
  The GVHD prophylaxis will consist of the following:
  * Cyclosporine on Day -3 to Day +100, maintaining a level of 250-500 ng/mL, then taper to Day +180.
  * Methylprednisolone 2 mg/kg/day on Day -2 and -1, 1 mg/kg/day on Day 0 to Day +28, then taper over 1 month. Oral prednisone may be substituted starting on Day 0 (1.2 mg/kg/day)
Period: Overall Study
Arm/Group | Hematopoietic Stem Cell Transplant
Started | 47
Completed | 46
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- Hemophagocytic Lymphohistiocytosis (HLH): Participants with Hemophagocytic Lymphohistiocytosis
- Other Primary Immune Deficiencies (PID): Participants with other primary immune deficiencies, including chronic active EBV disease, chronic granulomatous disease, hyper-immunoglobulin M syndrome, and immune dysregulation, polyendocrinopathy, enteropathy and X-linked (IPEX) syndrome
- Total: Total of all reporting groups
Arm/Group | Hemophagocytic Lymphohistiocytosis (HLH) | Other Primary Immune Deficiencies (PID) | Total
Number analyzed (Participants) | 34 | 12 | 46
Age, Customized [Count of Participants; unit: Participants]
  0-9 Years | 26 | 8 | 34
  10-19 Years | 7 | 2 | 9
  20-29 Years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 15
  Male | 23 | 8 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 26 | 9 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Karnofsky Performance Score (KPS) [Count of Participants; unit: Participants] — KPS describes patient-perceived global quality of life and functioning on a scale of 0-100.
  100: No evidence of disease; 90: Normal activity. Minor signs or symptoms of disease; 80: Normal activity with effort. Some signs or symptoms of disease; 70: Cares for self. Unable to continue normal activity; 60: Needs occasional assistance, but cares for most personal needs; 50: Needs considerable assistance and medical care; 40: Disabled. Needs special care and assistance; 30: Severely disabled. Hospital admission indicated; 20: Very sick. Active supportive therapy needed; 10: Moribund; 0: Dead
  Participants
    90-100 | 24 | 10 | 34
    80 | 6 | 2 | 8
    70 | 2 | 0 | 2
    60 | 1 | 0 | 1
    50 | 1 | 0 | 1
Primary Immune Deficiency Type [Count of Participants; unit: Participants] — Population: Participants with Primary Immune Deficiencies
  Participants
    number analyzed (Participants) | 0 | 12 | 12
    Chronic Active Epstein-Barr Virus |  | 3 | 3
    Chronic Granulomatous Disease |  | 5 | 5
    Hyperimmunoglobulin M Syndrome |  | 2 | 2
    IPEX |  | 2 | 2
Donor Type [Count of Participants; unit: Participants] — HLA matching and relatedness of donor to recipient
  Participants
    HLA Matched Sibling | 7 | 0 | 7
    1 HLA Locus Mismatched Relative | 0 | 1 | 1
    HLA Matched Unrelated | 16 | 9 | 25
    1 HLA Locus Mismatched Unrelated | 11 | 2 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Survival (OS)
Description: Overall survival is defined as survival of death from any cause.
Time Frame: 1 year and 18 months post-transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 46
percentage of participants
  1 year OS | 80.4 [68.6 to 88.2]
  18 month OS | 66.7 [52.9 to 77.3]

2. Secondary Outcome: Percentage of Participants With Overall Survival (OS) by Disease Type
Description: Overall survival is defined as survival of death from any cause.
Time Frame: 1 year and 18 months post-transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hemophagocytic Lymphohistiocytosis (HLH) | Other Primary Immune Deficiencies (PID)
Number analyzed (Participants) | 34 | 12
percentage of participants
  1 year OS | 82.4 [68.4 to 90.6] | 75.0 [47.4 to 89.5]
  18 month OS | 68.0 [51.8 to 79.7] | 62.5 [32.7 to 82.0]

3. Secondary Outcome: Percentage of HLH Participants With HLH Reactivation Post-Transplant
Description: Systemic HLH Reactivation: Post-transplant HLH reactivation is defined by clinical and lab evidence of pathologic inflammation (persistent fever, progressive cytopenias, rising ferritin and soluble IL2Rα, decreasing fibrinogen, hepatosplenomegaly, end-organ damage) not attributable to other causes.
  Central nervous system (CNS) HLH Reactivation: Reactivation of CNS inflammation in patients with HLH may present with or without altered mental status and is defined by pleocytosis in Cerebrospinal fluid (CSF) or an MRI consistent with CNS inflammation not attributable to other causes.
Time Frame: 1 year post-transplant
Population: Participants with HLH
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 34
percentage of participants | 14.7 [5.2 to 28.7]

4. Secondary Outcome: Percentage of Participants With Neutrophil Engraftment
Description: Time to absolute neutrophil count (ANC) engraftment is defined as the first of three measurements on different days that the patient has an absolute neutrophil count of ≥ 500x10^6/liter following conditioning regimen induced nadir.
Time Frame: Day 42 post-transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 46
percentage of participants | 100.0 [90.8 to 100.0]

5. Secondary Outcome: Percentage of Participants With Platelet Engraftment
Description: Platelet engraftment is defined as the first day of a minimum of three measurements on different days that the patient has achieved a platelet count > 20,000 / microliter AND the patient is platelet transfusion independent for a minimum of seven days following conditioning regimen induced nadir.
Time Frame: Day 100 post-transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 46
percentage of participants | 88.9 [73.3 to 95.6]

6. Secondary Outcome: Percentage of Participants Alive With Sustained Engraftment
Description: Sustained engraftment is defined as the occurrence of whole blood donor chimerism > 5% by Day 42 accompanied by the absence of any primary or secondary graft failure. Primary graft failure is defined as < 5% donor chimerism by Day +42, second stem cell infusion, DLI (except in the case of donor CTLs given for infection control), or second HCT following original HCT. Secondary graft failure is defined as < 5% donor chimerism following initial engraftment.
Time Frame: 1 year post-transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 46
percentage of participants | 39.1 [25.1 to 54.6]

7. Secondary Outcome: Percentage of Participants Alive With Sustained Engraftment by Disease Type
Description: as for outcome 6
Time Frame: 1 year post-transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hemophagocytic Lymphohistiocytosis (HLH) | Other Primary Immune Deficiencies (PID)
Number analyzed (Participants) | 34 | 12
percentage of participants | 41.2 [24.7 to 59.3] | 33.3 [9.9 to 65.1]

8. Secondary Outcome: Number of Participants With Acute Graft-Versus-Host Disease (GVHD)
Description: Acute GVHD is graded according to the scoring system proposed by Przepiorka et al.1995:
  Skin stage:
  0: No rash
  1. Rash <25% of body surface area
  2. Rash on 25-50% of body surface area
  3. Rash on > 50% of body surface area
  4. Generalized erythroderma with bullous formation
  Liver stage (based on bilirubin level)*:
  0: <2 mg/dL
  1. 2-3 mg/dL
  2. 3.01-6 mg/dL
  3. 6.01-15.0 mg/dL
  4. >15 mg/dL
  GI stage*:
  0: No diarrhea or diarrhea <500 mL/day
  1. Diarrhea 500-999 mL/day or persistent nausea with histologic evidence of GVHD
  2. Diarrhea 1000-1499 mL/day
  3. Diarrhea >1500 mL/day
  4. Severe abdominal pain with or without ileus * If multiple etiologies are listed for liver or GI, the organ system is downstaged by 1.
  GVHD grade:
  0: All organ stages 0 or GVHD not listed as an etiology I: Skin stage 1-2 and liver and GI stage 0 II: Skin stage 3 or liver or GI stage 1 III: Liver stage 2-3 or GI stage 2-4 IV: Skin or liver stage 4
Time Frame: 1 year post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 46
Participants
  Grade 0 or I | 35
  Grade II | 3
  Grade III | 5
  Grade IV | 3

9. Secondary Outcome: Percentage of Participants With Grade II-IV and Grade III-IV Acute GVHD
Description: as for outcome 8
Time Frame: Day 100 and 6 months post-transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 46
percentage of participants
  Grade II-IV Acute GVHD at Day 100 | 17.4 [8.1 to 29.7]
  Grade II-IV Acute GVHD at 6 Months | 26.1 [14.4 to 39.4]
  Grade III-IV Acute GVHD at Day 100 | 10.9 [4.0 to 21.3]
  Grade III-IV Acute GVHD at 6 Months | 17.4 [8.1 to 29.7]

10. Secondary Outcome: Number of Participants With Chronic GVHD
Description: Chronic GVHD is classified per 2005 NIH Consensus Criteria (Filipovich et al. 2005) into categories of severity: none, mild, moderate, and severe.
Time Frame: 1 year post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 46
Participants
  None | 34
  Mild | 10
  Severe | 2

11. Secondary Outcome: Percentage of Participants With Chronic GVHD
Description: Chronic GVHD is classified per 2005 NIH Consensus Criteria (Filipovich et al. 2005) into categories of severity: none, mild, moderate, and severe. Occurrence of chronic GVHD is defined as the occurrence of mild, moderate, or severe chronic GVHD per this classification.
Time Frame: 1 year post-transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 46
percentage of participants | 26.7 [14.6 to 40.4]

ADVERSE EVENTS:
Time Frame: 1 year post-transplant
Arm/Group | Hematopoietic Stem Cell Transplant
Serious Adverse Events (participants affected / at risk) | 14/46
Other Adverse Events (participants affected / at risk) | 0/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hematopoietic Stem Cell Transplant (N=46)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2)
Ventricular hypertrophy (Cardiac disorders) | 1 (1)
Death (General disorders) | 1 (1)
Serum sickness (Immune system disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Post transplant lymphoproliferative disorders (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypotension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-06-16): https://cdn.clinicaltrials.gov/large-docs/33/NCT01998633/Prot_SAP_ICF_000.pdf